CLINICAL TRIAL: NCT02026102
Title: A Pilot Trial of Patient Decision Aids for Implantable Cardioverter-Defibrillators (ICDs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 13-3152; 121483 (Other Grant/Funding Number: Patient Centered Outcomes Research Institute (PCORI))
Record Dates: First submitted 2013-12-12; First posted 2014-01-01 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Systolic Heart Failure; Sudden Cardiac Death
Keywords: decision aid; patient decision making; heart failure; ejection fraction; primary prevention; implantable cardioverter defibrillator; ICD; pilot trial; patient centered health care
MeSH Terms: conditions — Heart Failure, Systolic; Death, Sudden, Cardiac; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (No Intervention): Patients will receive no additional ICD specific information other than what is offered by the clinic consistent with usual care. The control group will be asked where they went for information in the follow-up interviews.
- ICD Decision Aid Toolkit (Experimental): In the intervention arm, research assistants will provide the patients with the toolkit of decision aids. At that time, participants will have the option of using all of the decision aids or just some of the decision aids. Participants who do not have access to the internet, will be offered a DVD (digital video disc) version of the video and they will be asked if they would like to arrange a visit where they can review the website with the research assistant.
  Interventions: Behavioral: ICD Decision Aid Toolkit

INTERVENTIONS:
Behavioral: ICD Decision Aid Toolkit — Research assistants will provide patients with a toolkit of decision aids. Participants will have the option of using all of the decision aids or just some of the decision aids.
  Arms: ICD Decision Aid Toolkit

SUMMARY:
The purpose of this study is to test the acceptability and feasibility of a "toolkit" of patient decision aids (PtDAs) for heart failure patients who are considering an ICD implant.

DETAILED DESCRIPTION:
Specific Aim 1: Examine acceptability and feasibility of a toolkit of patient decision aids (PtDAs) for patients with heart failure referred for primary prevention implantable cardioverter-defibrillators using a randomized control trial design across three diverse health care systems (Kaiser Colorado, The University of Colorado, and The Denver Veterans Hospital).

1. Measure the acceptability of the decision aids
2. Explore feasibility by measuring patient participation rates and adherence to the study protocol across all three sites.
3. Conduct a preliminary assessment of outcomes by measuring changes in decision quality (knowledge and value concordance), quality of life, depressive symptoms, health status, and spiritual well-being.

Specific Aim 2: Determine the relative value of the various tools in the toolkit through in-depth interviews from study participants and providers at each intervention site

ELIGIBILITY:
Inclusion Criteria:

* systolic heart failure (defined as an ejection fraction less than 35%)
* have been referred for a primary prevention ICD
* Note: Patients referred for an ICD with cardiac resynchronization therapy are NOT excluded.

Exclusion Criteria:

* Already have an ICD
* Non-English speaking (as the tools we have developed are only available in English currently)
* Other ICD indications (e.g. secondary prevention, hypertrophic obstructive cardiomyopathy)
* Cognitive Impairment defined only as people with an inability to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measure the acceptability and feasibility of the decision aids | pre-ICD discussion - baseline
  Acceptability-measure decision aid acceptability using modified version of decision aid acceptability developed by Barry et al.
  Feasibility-explore participation rates and adherence to study protocol; weekly team meetings to discuss recruitment strategies Knowledge: 21 item knowledge measure developed in-house Decision Conflict: validated 15-item decision conflict measure developed by O'Connor et al.
  Decision Regret: validated 5-item decision regret scale Decision choice: ultimate choice patient made about getting an ICD Decision participation: Prior to intervention, we measure patients' preferred role in decision making using the control preferences scale. After the decision, we measure the participants' actual role in decision making.
  Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS). Chart Review Outcome: For those that had not yet had a procedure, we will review the charts at the end of study to determine if they received an ICD or not.

SECONDARY OUTCOMES:
Determine relative value of the four decision aids | 3 months after baseline interview
  Determine the relative value of the various tools in the toolkit through in-depth interviews from study participants and providers at each intervention site.
  We will ask participants the following questions:
  * Have you made a decision about getting or not getting the ICD?
  * What information did you use to make your decision?
  * How are you feeling about your decision?
  * What else would have been helpful in making your decision?
  * (Intervention only) Did you use any of the decision aids you were given?
  * If yes, please tell us how you used them? Did the decision aids make you feel better or worse about your decision? Did you like one of them better than the others? Is there any aspect that wasn't helpful?
  * If no, please tell us why not? What would have been helpful?
  * Do you have any advice on the best way to deliver these decision aids to future patients?
Measure the acceptability and feasibility of the decision aids | within 4 weeks of meeting with electrophysiologist
  Acceptability-measure decision aid acceptability using modified version of decision aid acceptability developed by Barry et al.
  Feasibility-explore participation rates and adherence to study protocol; weekly team meetings to discuss recruitment strategies Knowledge: 21 item knowledge measure developed in-house Decision Conflict: validated 15-item decision conflict measure developed by O'Connor et al.
  Decision Regret: validated 5-item decision regret scale Decision choice: ultimate choice patient made about getting an ICD Decision participation: Prior to intervention, we measure patients' preferred role in decision making using the control preferences scale. After the decision, we measure the participants' actual role in decision making.
  Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS). Chart Review Outcome: For those that had not yet had a procedure, we will review the charts at the end of study to determine if they received an ICD or not.
Measure the acceptability and feasibility of the decision aids | 3 months after baseline interview
  Acceptability-measure decision aid acceptability using modified version of decision aid acceptability developed by Barry et al.
  Feasibility-explore participation rates and adherence to study protocol; weekly team meetings to discuss recruitment strategies Knowledge: 21 item knowledge measure developed in-house Decision Conflict: validated 15-item decision conflict measure developed by O'Connor et al.
  Decision Regret: validated 5-item decision regret scale Decision choice: ultimate choice patient made about getting an ICD Decision participation: Prior to intervention, we measure patients' preferred role in decision making using the control preferences scale. After the decision, we measure the participants' actual role in decision making.
  Anxiety and Depression: Hospital Anxiety and Depression Scale (HADS). Chart Review Outcome: For those that had not yet had a procedure, we will review the charts at the end of study to determine if they received an ICD or not.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel D Matlock, MD, MPH, Principal Investigator — University of Colorado, Denver
Locations (3):
- United States (3):
  - University of Colorado Hospital (UCH), Aurora, Colorado
  - Kaiser Permanente of Colorado, Denver, Colorado
  - Denver VA Medical Center, Denver, Colorado

REFERENCES:
- [Background] O'Connor AM, Wennberg JE, Legare F, Llewellyn-Thomas HA, Moulton BW, Sepucha KR, Sodano AG, King JS. Toward the 'tipping point': decision aids and informed patient choice. Health Aff (Millwood). 2007 May-Jun;26(3):716-25. doi: 10.1377/hlthaff.26.3.716. PMID 17485749
- [Background] O'Connor AM, Bennett CL, Stacey D, Barry M, Col NF, Eden KB, Entwistle VA, Fiset V, Holmes-Rovner M, Khangura S, Llewellyn-Thomas H, Rovner D. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2009 Jul 8;(3):CD001431. doi: 10.1002/14651858.CD001431.pub2. PMID 19588325
- [Background] Volandes AE, Paasche-Orlow MK, Barry MJ, Gillick MR, Minaker KL, Chang Y, Cook EF, Abbo ED, El-Jawahri A, Mitchell SL. Video decision support tool for advance care planning in dementia: randomised controlled trial. BMJ. 2009 May 28;338:b2159. doi: 10.1136/bmj.b2159. PMID 19477893
- [Background] Col NF, Ngo L, Fortin JM, Goldberg RJ, O'Connor AM. Can computerized decision support help patients make complex treatment decisions? A randomized controlled trial of an individualized menopause decision aid. Med Decis Making. 2007 Sep-Oct;27(5):585-98. doi: 10.1177/0272989X07306781. Epub 2007 Sep 14. PMID 17873260
- [Background] Jibaja-Weiss ML, Volk RJ, Granchi TS, Neff NE, Robinson EK, Spann SJ, Aoki N, Friedman LC, Beck JR. Entertainment education for breast cancer surgery decisions: a randomized trial among patients with low health literacy. Patient Educ Couns. 2011 Jul;84(1):41-8. doi: 10.1016/j.pec.2010.06.009. Epub 2010 Jul 7. PMID 20609546
- [Background] Stevenson LW, Desai AS. Selecting patients for discussion of the ICD as primary prevention for sudden death in heart failure. J Card Fail. 2006 Aug;12(6):407-12. doi: 10.1016/j.cardfail.2006.06.001. PMID 16911905
- [Background] Bardy GH, Lee KL, Mark DB, Poole JE, Packer DL, Boineau R, Domanski M, Troutman C, Anderson J, Johnson G, McNulty SE, Clapp-Channing N, Davidson-Ray LD, Fraulo ES, Fishbein DP, Luceri RM, Ip JH; Sudden Cardiac Death in Heart Failure Trial (SCD-HeFT) Investigators. Amiodarone or an implantable cardioverter-defibrillator for congestive heart failure. N Engl J Med. 2005 Jan 20;352(3):225-37. doi: 10.1056/NEJMoa043399. PMID 15659722
- [Background] Bristow MR, Saxon LA, Boehmer J, Krueger S, Kass DA, De Marco T, Carson P, DiCarlo L, DeMets D, White BG, DeVries DW, Feldman AM; Comparison of Medical Therapy, Pacing, and Defibrillation in Heart Failure (COMPANION) Investigators. Cardiac-resynchronization therapy with or without an implantable defibrillator in advanced chronic heart failure. N Engl J Med. 2004 May 20;350(21):2140-50. doi: 10.1056/NEJMoa032423. PMID 15152059
- [Background] Moss AJ, Zareba W, Hall WJ, Klein H, Wilber DJ, Cannom DS, Daubert JP, Higgins SL, Brown MW, Andrews ML; Multicenter Automatic Defibrillator Implantation Trial II Investigators. Prophylactic implantation of a defibrillator in patients with myocardial infarction and reduced ejection fraction. N Engl J Med. 2002 Mar 21;346(12):877-83. doi: 10.1056/NEJMoa013474. Epub 2002 Mar 19. PMID 11907286
- [Background] Kadish A, Dyer A, Daubert JP, Quigg R, Estes NA, Anderson KP, Calkins H, Hoch D, Goldberger J, Shalaby A, Sanders WE, Schaechter A, Levine JH; Defibrillators in Non-Ischemic Cardiomyopathy Treatment Evaluation (DEFINITE) Investigators. Prophylactic defibrillator implantation in patients with nonischemic dilated cardiomyopathy. N Engl J Med. 2004 May 20;350(21):2151-8. doi: 10.1056/NEJMoa033088. PMID 15152060
- [Background] Goldenberg I, Moss AJ, Hall WJ, McNitt S, Zareba W, Andrews ML, Cannom DS; Multicenter Automatic Defibrillator Implantation Trial (MADIT) II Investigators. Causes and consequences of heart failure after prophylactic implantation of a defibrillator in the multicenter automatic defibrillator implantation trial II. Circulation. 2006 Jun 20;113(24):2810-7. doi: 10.1161/CIRCULATIONAHA.105.577262. Epub 2006 Jun 12. PMID 16769917
- [Background] Noyes K, Corona E, Zwanziger J, Hall WJ, Zhao H, Wang H, Moss AJ, Dick AW; Multicenter Automatic Defibrillator Implantation Trial II. Health-related quality of life consequences of implantable cardioverter defibrillators: results from MADIT II. Med Care. 2007 May;45(5):377-85. doi: 10.1097/01.mlr.0000257142.12600.c1. PMID 17446823
- [Background] Mark DB, Anstrom KJ, Sun JL, Clapp-Channing NE, Tsiatis AA, Davidson-Ray L, Lee KL, Bardy GH; Sudden Cardiac Death in Heart Failure Trial Investigators. Quality of life with defibrillator therapy or amiodarone in heart failure. N Engl J Med. 2008 Sep 4;359(10):999-1008. doi: 10.1056/NEJMoa0706719. PMID 18768943
- See also: Decision Aid for Heart Failure Patients Considering an Implantable Cardioverter Defibrillator — https://www.patientdecisionaid.org/